CLINICAL TRIAL: NCT02588742
Title: The Effect of Melatonin on Postoperative Delirium in Elderly ICU Patients : Randomized, Placebo-controlled, Double Blind Study
Brief Title: The Effect of Melatonin on Postoperative Delirium in Elderly ICU Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminate the study because it is difficult to recruit the subject.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2014-1038
Record Dates: First submitted 2015-10-19; First posted 2015-10-28 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-02

CONDITIONS: Delirium
Keywords: elderly ICU patients
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- melatonin group (Experimental): Patients in the melatonin group are given 5mg of melatonin at 8 pm the day before surgery, POD#0, POD#1, POD#2, POD#3, POD#4, and POD#5.
  Interventions: Dietary Supplement: Melatonin
- control group (Placebo Comparator): Patients in the control group are given placebo at 8 pm the day before surgery, POD#0, POD#1, POD#2, POD#3, POD#4, and POD#5.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Patients in the melatonin group are given 5mg of melatonin at 8 pm the day before surgery, POD#0, POD#1, POD#2, POD#3, POD#4, and POD#5.
  Arms: melatonin group
Dietary Supplement: Placebo — Patients in the control group are given placebo at 8 pm the day before surgery, POD#0, POD#1, POD#2, POD#3, POD#4, and POD#5.
  Arms: control group

SUMMARY:
Delirium in older patients is associated with increased mortality and health care costs. And delirium is frequent in intensive care unit (ICU). Circadian rhythm alteration is one of the most important risk factor for developing delirium. In this study, investigators will investigate the effect of administration of melatonin on postoperative delirium in elderly ICU patients.

Randomly selected patients of the melatonin group are given 5mg of melatonin in the evening from the day before surgery to the the 5th postoperation day. In contrast, patients in the control group are given placebo.

Primary outcome of this study is the incidence of postoperative delirium measured by ICD-SC (Intensive Care delirium Screening Checklist). And secondary outcome includes intra-procedural hemodynamics measured by amount of used vasopressors, heart rate and blood pressure, total amount of sedatives, total amount of analgesics, duration of mechanical ventilation, duration of ICU stay.

Thus, investigators perform this study to investigate the relationship between delirium and circadian rhythm.

ELIGIBILITY:
Inclusion Criteria:

* older than 50 years old
* patients who admitted to ICU after surgery

Exclusion Criteria:

* Subjects are ineligible if they have cognitive dysfunction,
* disabling mental change disorder,
* alcohol addiction,
* dementia,
* cerebrovascular accident,
* transient ischemic attack,
* carotid artery stenosis,
* autoimmune disease,
* patients who are unable to communicate or speak Korean,
* emergent operation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02-02; Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
incidence of delirium | 5 days after surgery
  The score of ICD-SC(Intensive Care Delirium Screening Checklist) will be recorded to identify the incidence of delirium for 5 days after surgery.

SECONDARY OUTCOMES:
change of amount of used vasopressors as a measure of intraoperative hemodynamics | up to 5 days
  intra-procedural hemodynamics measured by amount of used vasopressors
total amount of sedatives | up to 5 days
total amount of analgesics | up to 5 days
duration of mechanical ventilation | up to 5 days
duration of ICU stay | up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea